CLINICAL TRIAL: NCT03634605
Title: Assessment of Tetracycline Pleurodesis in Prevention of Primary Spontaneous Pneumothorax Recurrence in Patients With Normal CT-scan
Brief Title: Effect of Tetracycline Pleurodesis on Prevention of Primary Spontaneous Pneumothorax Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, Assistant professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 395351
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Primary Spontaneous Pneumothorax
Keywords: Tetracycline; Pleurodesis
MeSH Terms: conditions — Pneumothorax | interventions — Saline Solution; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case Group (Experimental): Chemical pleurodesis for the this group was done using 2 grams of tetracycline 3% ointment (Aerotex®, Sina Daru, Tehran, Iran), 5 milliliter of lidocaine 2% and 50 milliliter normal saline that was injected through embedded thoracostomy tube
  Interventions: Procedure: Chemical pleurodesis; Drug: Tetracycline Topical Ointment; Drug: Normal saline; Drug: Lidocaine 2% Injectable Solution
- Control Group (Placebo Comparator): Chemical pleurodesis for this group was done using 5 milliliter of lidocaine 2% and 50 milliliter normal saline that was injected through embedded thoracostomy tube
  Interventions: Procedure: Chemical pleurodesis; Drug: Normal saline; Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Procedure: Chemical pleurodesis
Drug: Tetracycline Topical Ointment
  Arms: Case Group
Drug: Normal saline
Drug: Lidocaine 2% Injectable Solution

SUMMARY:
Primary spontaneous pneumothorax (PSP) defines as presence of air in chest cavity occurs most commonly in young, tall, and smoker men without underlying lung disease.

Trends for PSP treatment tend toward more invasive procedures. Thoracotomy with pleurectomy and bullectomy is definitive treatment of PSP which significantly reduces recurrence probability. This procedure has been reported to cause high rate of morbidity and mortality. Thus video-assisted thoracoscopic surgery (VATS) has become the preferred method for treatment of PSP with recurrence rate of 5-10%. For persistent or recurrent cases, mechanical or chemical pleurodesis have been suggested.

Based on guidelines patients with large size of lesions in CT or with unstable condition should undergo surgical procedure for recurrence prevention but Patients with small lesion size and stable condition can be only observed. Conservative management of PSP is safe and effective, but as mentioned this method has high recurrence rate. On the other hand fear of recurrence can negatively affect patients' quality of life, so that some patients prefer surgical intervention to observation management. Also some studies recommend invasive treatments because of cost effectiveness of this methods.

As mentioned above, chemical pleurodesis is a usual method for treatment in patients with persistent or recurrent spontaneous pneumothorax. This method has been done using variety of chemical agents including tetracycline, minocycline, blood, and talc to irritate pleura. According to different studies tetracycline has the highest efficacy between irritant agents.

In current study, the investigators have aimed to assess tetracycline chemical pleurodesis through tube thoracostomy in prevention of spontaneous pneumothorax in symptom free patients with normal CT-scan following first episode of PSP.

ELIGIBILITY:
Inclusion Criteria:

* First episode of primary spontaneous pneumothorax
* Do not have bullae in CT-scan
* No history of chest trauma or thoracic surgery

Exclusion Criteria:

* History of chest trauma or thoracic surgery and start/quiting of smoking during past year.
* Not willing to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2016-10-22 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Recurrence | 12 months
  Evaluation of recurrence of primary spontaneous pneumothorax in 2 study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan Unviersity of medical Sciences, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No